CLINICAL TRIAL: NCT07371325
Title: Efficacy of Pediococcus Acidilactici as add-on to Antipsychotic Drugs on Metabolic Syndrome Disturbances in First-episode Psychosis and Schizophrenia Spectrum Disorders. A Double-blind Placebo-controlled Trial.
Acronym: GLUCOPSICO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Manuel Jesús Cuesta Zurita (Other)
Collaborators: GENBIOMA Aplicaciones SL (Unknown); Universidad Pública de Navarra (Other)
Responsible Party: Sponsor-Investigator, Manuel Jesús Cuesta Zurita, PSYCHIATRIST, Fundacion Miguel Servet
Organization: Fundacion Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: GLUCOPSICOBIOMICS_2025
Record Dates: First submitted 2026-01-08; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: SCHIZOPHRENIA 1 (Disorder); Metabolic Abnormalities; Postbiotic Supplement
Keywords: Schizophrenia; First-episode psychosis; Metabolic Syndrome; Postbiotic; Atypical antipsychotics
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: A double-blind placebo-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FEP and postbiotic (Experimental): Participants with FEP diagnostic taking postbiotic and atypical antipsychotics
  Interventions: Dietary Supplement: Pediococcus acidilactici, pA1c®HI postbiotic supplementation taking participants; Drug: Atypical antipsychotics (AAP)
- SSD and postbiotic (Experimental): Participants with SSD diagnostic taking postbiotic and atypical antipsychotics
  Interventions: Dietary Supplement: Pediococcus acidilactici, pA1c®HI postbiotic supplementation taking participants; Drug: Atypical antipsychotics (AAP)
- FEP and placebo (Placebo Comparator): Participants with FEP diagnostic taking placebo and atypical antipsychotics
  Interventions: Drug: Atypical antipsychotics (AAP)
- SSD and placebo (Placebo Comparator): Participants with SSD diagnostic taking placebo and atypical antipsychotics
  Interventions: Drug: Atypical antipsychotics (AAP)

INTERVENTIONS:
Dietary Supplement: Pediococcus acidilactici, pA1c®HI postbiotic supplementation taking participants — This study is the first study based on postbiotics instead of probiotics, pA1C®HI will be included as add on to the treatment with atypical antipsychotics in patients diagnosed with FEP or SSD. We include in our study the monitoring of glucose levels by means of sensors that will allow not only the recording of these average daily and weekly glucose levels but also the physical activity performed by the participant along the whole study. We also analyze the microbiota, responsible for metabolic functions, through metatranscriptome of intestinal microbiota from faecal samples from participants
  Arms: FEP and postbiotic; SSD and postbiotic
Drug: Atypical antipsychotics (AAP) — This study participants will continue with their established drug treatment as prescribed by their referring therapists. In the event of any changes to the treatment, the appropriate record will be made.

SUMMARY:
The aim of the present study is to evaluate the effectiveness of the addition of the postbiotic Pediococcus acidilactici (pA1c®HI) on amelioration of metabolic disturbances in patients with (FEP) or (SSD) treated with antipsychotic drugs.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of an add-on postbiotic (Pediococcus acidilactici, pA1c®HI) to antipsychotic drugs on metabolic disturbances and psychopathological dimensions in patients diagnosed with first episode psychotic (FEP) or schizophrenia spectrum disorder (SSD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PEP or TEESQ, according to DSM 5 criteria, aged between 18 and 65 years
* Having received antipsychotic treatment for at least 8 weeks before starting the study

Exclusion Criteria:

* Inability to give informed consent, lack of a representative or legal guardian capable of giving consent
* Intellectual disability
* Clinically significant medical condition (congestive heart failure, liver disease, renal failure, acute pancreatitis, cancer undergoing active treatment, HIV, or other immunodeficiency)
* Active substance use in the last 3 months (except nicotine)
* Antibiotic medication in the previous 14 days
* Celiac disease
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-09-08 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12).
  1. Total cholesterol
  Description: Measurement of total cholesterol in the blood. Includes LDL, HDL, and other fractions. It is a general marker of cardiovascular risk.
  Units: mg/dL
  Ranges:
  Desirable: < 200 mg/dL
  High limit: 200-239 mg/dL
  High: ≥ 240 mg/dL
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12)
  2. LDL cholesterol (Low-Density Lipoprotein)
  Description: Known as "bad cholesterol." High levels are associated with atherosclerosis and cardiovascular disease.
  Units: mg/dL
  Ranges:
  Optimal: < 100 mg/dL
  Near optimal: 100-129 mg/dL
  High limit: 130-159 mg/dL
  High: 160-189 mg/dL
  Very high: ≥ 190 mg/dL
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12)
  3. HDL cholesterol (High-Density Lipoprotein)
  Description: Known as "good cholesterol." Helps remove cholesterol from the arteries.
  Units: mg/dL
  Ranges:
  Low (cardiovascular risk):
  Men: < 40 mg/dL
  Women: < 50 mg/dL
  Adequate/protective: ≥ 60 mg/dL
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12)
  4. Triglycerides
  Description: Type of fat in the blood related to energy metabolism. High values are associated with metabolic syndrome and cardiovascular risk.
  Units: mg/dL
  Ranges (fasting):
  Normal: < 150 mg/dL
  High limit: 150-199 mg/dL
  High: 200-499 mg/dL
  Very high: ≥ 500 mg/dL
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12)
  5. Plasma glucose
  Description: Blood glucose concentration, a key indicator of carbohydrate metabolism.
  Units: mg/dL
  Ranges (fasting):
  Normal: 70-99 mg/dL
  Impaired fasting glucose (prediabetes): 100-125 mg/dL
  Diabetes: ≥ 126 mg/dL
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12)
  6. Insulin
  Description: Hormone produced by the pancreas that regulates glucose uptake by tissues.
  Units: µU/mL (or mIU/L)
  Ranges (fasting):
  Approximate normal: 2-25 µU/mL
  Elevated values may suggest insulin resistance.
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12)
  7. Glycosylated hemoglobin (HbA1c)
  Description: Reflects the average blood glucose level over the past 2-3 months.
  Units: %
  Ranges:
  Normal: < 5.7%
  Prediabetes: 5.7-6.4%
  Diabetes: ≥ 6.5%
Metabolic Disturbances | Beginning (week 0) and end of the study (week 12)
  8. HOMA-R (or HOMA-IR)
  Description: Index that estimates insulin resistance, calculated from fasting glucose and insulin.
  Formula:
  HOMA-IR = Insulin (µU/mL) × Glucose (mg/dL) / 405
  Units: No units (index)
  Guideline ranges:
  Normal: < 2.0
  Mild insulin resistance: 2.0-2.9
  Significant insulin resistance: ≥ 3.0

SECONDARY OUTCOMES:
Clinical Measures | Along the study: week 0, week 6, and week 12
  Positive and Negative Symptoms
  1. Positive and Negative Syndrome Scale (PANSS)
  Description: A widely used clinical scale for assessing the severity of positive and negative symptoms and general psychopathology in schizophrenia and other psychotic disorders.
  Structure: 30 items divided into:
  Positive subscale (7 items)
  Negative subscale (7 items)
  General psychopathology (16 items)
  Scoring: Each item is scored from 1 (absent) to 7 (extreme).
  Ranges:
  Total score: 30-210
  The higher the score, the greater the symptom severity.
  Guideline interpretation (total):
  Mild: ~58-75
  Moderate: ~75-95
  Severe: >95
Clinical Measures | Along the study: week 0, week 6, and week 12
  2. Brief Negative Symptoms Scale (BNSS)
  Description: Instrument designed specifically to assess negative symptoms in detail.
  Domains assessed (6):
  Anhedonia
  Asociality
  Avolition
  Affective flattening
  Alogia
  Lack of emotional distress
  Structure: 13 items
  Scoring: Items scored from 0 (absent) to 6 (severe).
  Total range: 0-78
  Interpretation:
  Higher scores indicate greater severity of negative symptoms.
Clinical Measures | Along the study: week 0, week 6, and week 12
  Cognitive symptoms 3. Screening for Cognitive Impairment in Psychiatry (SCIP)
  Description: Brief test for detecting cognitive impairment in psychiatric patients.
  Domains assessed:
  Verbal learning
  Working memory
  Verbal fluency
  Processing speed
  Delayed memory
  Duration: ~15 minutes
  Scoring: Approximate total scale 0-100 (depending on version).
  Interpretation:
  Lower scores indicate greater cognitive impairment.
  Cut-off points adjusted for age and educational level are used.
Clinical measures | Along the study: week 0, week 6, and week 12
  4. MATRICS Consensus Cognitive Battery (MCCB)
  Description: Standardized reference battery for assessing cognition in schizophrenia.
  Domains assessed (7):
  Processing speed
  Attention/vigilance
  Working memory
  Verbal learning
  Visual learning
  Reasoning and problem solving
  Social cognition
  Score:
  T scores (mean = 50, SD = 10)
  Interpretation:
  T < 40: below-average performance
  T 40-60: normal range
  T > 60: above-average performance
Clinical Measures | Along the study: week 0, week 6, and week 12
  5. Cognitive Reserve Assessment Scale in Health (CRASH)
  Description: Scale designed to estimate cognitive reserve, considering premorbid and sociocultural factors.
  Areas assessed:
  Educational level
  Occupation
  Cognitive and leisure activities
  Premorbid intellectual level
  Score: Composite index (no units).
  Interpretation:
  Higher scores indicate greater cognitive reserve, associated with a better functional prognosis.
  Affective symptoms 6. Calgary Depression Scale for Schizophrenia (CDSS)
  Description: Specific scale for assessing depressive symptoms in patients with schizophrenia, differentiating them from negative or extrapyramidal symptoms.
  Structure: 9 items
  Scoring: Items from 0 (absent) to 3 (severe).
  Total range: 0-27
  Interpretation:
  ≥ 6 points suggests the presence of clinically significant depression.
Clinical Measures | Along the study: week 0, week 6, and week 12
  Motor symptoms 7. Simpson-Angus Scale (SAS)
  Description: Instrument for assessing extrapyramidal symptoms, especially antipsychotic-induced parkinsonism.
  Structure: 10 items
  Scoring: Items from 0 (normal) to 4 (severe).
  Total score: Average of items or total sum.
  Interpretation:
  Higher scores indicate greater severity of motor symptoms.
Clinical Measures | Along the study: week 0, week 6, and week 12
  Overall functioning 8. Global Assessment of Functioning Scale (GAF)
  Description: Global scale that assesses psychological, social, and occupational functioning.
  Range: 0-100
  Interpretation:
  91-100: superior functioning
  71-90: minimal symptoms
  51-70: mild symptoms
  31-50: severe symptoms
  ≤ 30: severe impairment of functioning
Anthropometric Parameters | Along the study: week 0, week 6, and week 12.
  1. Weight
  Description: Measurement of the individual's total body mass.
  Units: kilograms (kg)
  Reference ranges:
  There are no universal "normal" ranges, as weight must be interpreted in relation to height, sex, and body composition. It is mainly used to calculate BMI.
Anthropometric Parameters | Along the study: week 0, week 6, and week 12
  2. Height
  Description: Body length measured in an upright position, from the soles of the feet to the top of the head.
  Units: centimeters (cm) or meters (m)
  Reference ranges:
  Variable depending on sex, age, and ethnicity; used primarily to calculate BMI.
Anthropometric Parameters | Along the study: week 0, week 6, and week 12
  3. Body Mass Index (BMI)
  Description: Indirect indicator of body fat that relates weight to height.
  Formula:
  BMI = weight (kg)/height (m)2
  Units: kg/m²
  Ranges (WHO):
  Underweight: < 18.5 kg/m²
  Normal weight: 18.5-24.9 kg/m²
  Overweight: 25.0-29.9 kg/m²
  Grade I obesity: 30.0-34.9 kg/m²
  Obesity grade II: 35.0-39.9 kg/m²
  Obesity grade III: ≥ 40 kg/m²
Anthropometric Parameters | Along the study: week 0, week 6, and week 12
  4. Waist circumference
  Description: Measurement of abdominal circumference, used as an indicator of visceral fat and cardiometabolic risk.
  Units: centimeters (cm)
  Cut-off points (cardiometabolic risk):
  Men: ≥ 102 cm
  Women: ≥ 88 cm (Some European criteria use ≥94 cm in men)
Anthropometric Parameters | Along the study: week 0, week 6, and week 12
  5. Heart rate
  Description: Number of heartbeats per minute at rest.
  Units: beats per minute (bpm)
  Ranges (resting, adults):
  Normal: 60-100 bpm
  Bradycardia: < 60 bpm
  Tachycardia: > 100 bpm
Anthropometric Parameters | Along the study: week 0, week 6, and week 12
  6. Blood pressure
  Description: Force exerted by blood against arterial walls, expressed as systolic/diastolic pressure.
  Units: millimeters of mercury (mmHg)
  Ranges (clinical guidelines):
  Normal: < 120 / < 80 mmHg
  Elevated: 120-129 / < 80 mmHg
  Grade 1 hypertension: 130-139 / 80-89 mmHg
  Grade 2 hypertension: ≥ 140 / ≥ 90 mmHg
Anthropometric Parameters | Along the study: week 0, week 6, and week 12
  7. Skin folds (Skinfold thickness)
  Description: Measurement of subcutaneous adipose tissue thickness using a skinfold caliper; allows estimation of body fat percentage.
  Units: millimeters (mm)
  Common measurement sites:
  Triceps
  Subscapular
  Suprailiac
  Abdominal
  Thigh
  Reference ranges:
  There are no universal values; results are interpreted:
  By summing skinfolds
  By applying predictive equations (e.g., Durnin-Womersley, Jackson-Pollock)
  Interpretation:
  Higher values indicate greater subcutaneous adiposity.

CONTACTS AND LOCATIONS:
Locations (1):
- Navarrabiomed, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang, D., Zhang, F., Yang, Y., Liu, C., Xiao, J., Long, Y., Huang, J., Peng, X., Wang, W., Wang, X., Davis, J. M., Zhao, J., & Wu, R. (2021). Probiotic supplements reduce antipsychotic-induced metabolic disturbances in drug-naïve first-episode schizophrenia. https://doi.org/10.1101/2021.02.16.21251872
- [Background] Pillinger, T., McCutcheon, R. A., Vano, L., Mizuno, Y., Arumuham, A., Hindley, G., Beck, K., Natesan, S., Efthimiou, O., Cipriani, A., & Howes, O. D. (2020). Comparative effects of 18 antipsychotics on metabolic function in patients with schizophrenia, predictors of metabolic dysregulation, and association with psychopathology: a systematic review and network meta-analysis. The Lancet Psychiatry, 7(1), 64-77. https://doi.org/10.1016/S2215-0366(19)30416-X
- [Background] Tomasik, J., Lago, S. G., Vázquez-Bourgon, J., Papiol, S., Suárez-Pinilla, P., Crespo-Facorro, B., & Bahn, S. (2019). Association of Insulin Resistance With Schizophrenia Polygenic Risk Score and Response to Antipsychotic Treatment. JAMA Psychiatry, 76(8), 864. https://doi.org/10.1001/jamapsychiatry.2019.0304
- [Background] Yavorov-Dayliev, D., Milagro, F. I., Ayo, J., Oneca, M., & Aranaz, P. (2022). Pediococcus acidilactici CECT9879 (pA1c) Counteracts the Effect of a High-Glucose Exposure in C. elegans by Affecting the Insulin Signaling Pathway (IIS). International Journal of Molecular Sciences, 23(5), 2689. https://doi.org/10.3390/ijms23052689